CLINICAL TRIAL: NCT03784118
Title: Study on Complications After Arterial Line Placement and the Risk Factors in Children
Brief Title: Complications Associated with Arterial Line Placement in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H1812-032-991
Record Dates: First submitted 2018-12-11; First posted 2018-12-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Complications After Arterial Catheterization
MeSH Terms: interventions — Ultrasonography; Perfusion Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children (Experimental): Children who are followed up after arterial catheterization for evaluation of complications, using ultrasonography
  Interventions: Diagnostic Test: Ultrasonography; Diagnostic Test: perfusion index

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Ultrasonography is used to evaluate the change in artery size after arterial catheterization and to assess the complication in children
Diagnostic Test: perfusion index — measurement of perfusion index immediately after arterial catheterization until surgery end, in arterial catheterization site and contralateral site.

SUMMARY:
The purpose of this study is to find the risk factors for complications following arterial line catheterization. Ultrasonography is used to evaluate the size of artery which is cannulated, before and after catheterization. The complications include ischemia, bleeding, thrombosis and so on.

DETAILED DESCRIPTION:
artery observation with ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under 5 years of age who require invasive arterial pressure monitoring

Exclusion Criteria:

* Patients who do not need invasive arterial pressure monitoring

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence of complications associated with arterial catheterization | within 5 days after arterial catheterization
  Number of participants with complications following arterial catheterization. The complications include thrombus, ischemia, oozing or bleeding, and color change, etc. If any of these occur, it is assumed that complications have occurred.

SECONDARY OUTCOMES:
Time-dependent changes in perfusion index | from arterial catheterization to the end of surgery
  Perfusion index was continuously monitored throughout surgery, on both sides: the digit on the side of the arterial line placement and the opposite side
Age as a risk factor | within 5 days after arterial catheterization
  To evaluate the age as one of the risk factors for complications following arterial catheterization using univariable logistic regression analysis.
Number of attempts as a risk factor | within 5 days after arterial catheterization
  To evaluate the number of attempts of arterial catheterization as one of the risk factors for complications
Duration of catheterization as a risk factor | within 5 days after arterial catheterization
  To evaluate the duration of catheterization as one of the risk factors for complications

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JH, Park JB, Ji SH, Jang YE, Kim EH, Kim JT, Kim HS. Immediate complications and risk factors following radial arterial catheterisation in paediatric patients at a tertiary centre. Eur J Anaesthesiol. 2025 Sep 8. doi: 10.1097/EJA.0000000000002268. Online ahead of print. PMID 40923190